CLINICAL TRIAL: NCT06406179
Title: Randomized Controlled Multicenter Trial to Evaluate the Efficacy and Safety of Dd-cfDNA in Routine Patient Care in Kidney Transplant Recipients
Brief Title: Evaluation of the Efficacy of Dd-cfDNA in Routine Patient Care in Kidney Transplant Recipients"
Acronym: AI-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP231641
Record Dates: First submitted 2024-04-29; First posted 2024-05-09 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Renal Transplantation
Keywords: renal transplantation rejection; non-invasive biomarker (dd-cfDNA ); risk evaluation; randomized trial; Gene expression

STUDY DESIGN:
Intervention Model Description: This is a 18-months follow-up national, multicenter, prospective , randomized, biomarker strategy design trial, whereby kidney transplant patients will be randomized 1:1 at the time of transplantation in 2 study groups.
  * Group I ("routine group"): during the first 18 months after transplantation, patients will follow a standard clinical follow-up based on kidney allograft function (serum creatinine, estimated glomerular filtration rate (eGFR), proteinuria). Allograft biopsies will be performed according the clinical practice of the center and the medical decision during the visits at M3, M12 or for clinical indication (CI).
  * Group II ("dd-cfDNA-guided"): As in the routine group at M3, M12 and at CI visits, patients will have clinical follow-up based on the investigators' routines. In addition, physicians will receive a report containing dd-cfDNA results and relevant medical parameters to help them decide whether or not to perform a biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I : routine group (No Intervention): patients will follow a standard clinical follow-up based on kidney allograft function (serum creatinine, estimated glomerular filtration rate (eGFR), proteinuria) and a surveillance allograft biopsy performed at 3 and 12 months after transplantation (M3 and M12) and for clinical indication whenever considered necessary by the clinician (CI), on the basis of 5 CI visits maximum expected per patient between D0 and M18. The standard of care comprises two biopsy cores: one is dedicated to histology. The paraffin-embedded core dedicated to SOC histology will be used for gene expression profiling and digital pathology imaging after SOC procedures .
- Group II: dd-cfDNA-guided (Experimental): Patients will follow a dd-cfDNA-guided strategy based on dd-cfDNA levels in the blood associated with relevant clinical data on the basis of its detection and prediction capacities for rejection at M3, M12 and during visits for clinical indication (5 CI visits maximum expected per patient between D0 and M18 to decide whether a biopsy is performed within the first 18 months of follow-up.
  Patients will be classified in "High risk" and "Low risk" depending on the dd-cfDNA integrative report generated by PARCC INSERM UMR 970 after centralization of dd-cfDNA results.
  If the patient is stratified into the "high-risk of rejection" subgroup, they can decide to perform the biopsy. In any case, the decision to perform the biopsy is left to the appreciation of the physician. They will report their awareness of the report's result to guide the act of biopsy in the eCRF.
  like in Group I, the standard of care comprises two biopsy cores
  Interventions: Biological: dd-cfDNA-guided

INTERVENTIONS:
Biological: dd-cfDNA-guided — In groups I and II, the blood sample for dd-cfDNA assay will be taken on D0, just prior to transplantation, for all patients.
  in addition, for patients following a dd-cf DNA-guided strategy based on dd-cf DNA ; samples for dd-cf DNA assay will be taken at M3 and M12 visits and at visits for clinical indication (5 maximum) and the blood will be sent to the PARCC technical platform of INSERM UMR 970. By combining the dd-cfDNA level and relevant medical data, an integration report will be sent to the centers to stratify patients into high-risk or low-risk rejection profiles.
  If the patient is classified in the "low risk of rejection" subgroup, he may decide not to perform the biopsy. If the patient is classified in the "high risk of rejection" subgroup, he may decide to perform the biopsy within 15 days of the sample being taken. the decision to perform the biopsy is left to the discretion of the physician.
  Arms: Group II: dd-cfDNA-guided

SUMMARY:
The investigator hypothesizes that the combined use of (1) Donor-derived cell-free DNA (dd-cfDNA) in peripheral blood predicting anti-donor immunological activation or quiescence (2) interactive and actionable data analytics delivered at the bedside will promote safe clinical follow-up of kidney transplant patients with less need for invasive biopsy and less induced risk surveillance by allograft protocol biopsies to assess allograft rejection in clinically stable kidney transplant patients.

In addition, the evaluation of the transcriptional changes in tissue samples in selected patients using automated processing of digital slide images and intragraft gene expression profiles will provide a better diagnosis of the rejection mechanisms to provide the best therapeutic approach as compared to current clinical practice.

We therefore propose a French, multicenter, prospective randomized trial comparing two strategies of follow-up: in the first group, a biopsy is performed at M3, M12 and for clinical indication whenever considered necessary by the clinician during the first 18 months of follow-up after transplant. In the second group, patients will have the same follow-up as in the first group, but reports providing dd-cfDNA results and relevant medical parameters will be provided to the physician to help him in the decision to perform a biopsy or not.

DETAILED DESCRIPTION:
The main objective of the study is to assess whether the use of donor-derived cell-free DNA (dd-cfDNA) as an immunological biomarker combined with clinical data to decrease the number of allograft biopsies during the first 18 months after transplantation.

500 new transplanted patients in 6 French clinical transplant sites will be included in the prospective multicenter AI-CARE trial. Recruitment of patients will start on the day of transplantation (or 8 days before for transplantations with living donor) and data/samples collected at 3 months and 12 months after transplantation and during visits for clinical indication within the first 18 months of follow-up. Realization of all the acts for the research are representing the usual medical practice (Standard Of Care: SOC) except one additional blood sample for dd-cfDNA analyses that will be collected and analyzed specifically for the research. The paraffin-embedded core dedicated to SOC histology will be used for gene expression profiling and digital pathology imaging after SOC procedures.

Using the newest information derived from dd-cfDNA analyses combined with clinical data, dd-cfDNA will allow us to identify kidney transplant patients at low- and high-risk of rejection.

using non-invasive dd-cfDNA levels combined with clinical data, preventing unnecessary allograft biopsies which are invasive, with and present a potential risk of complications for the patients and costly burden to the healthcare

ELIGIBILITY:
Inclusion Criteria:

* All men and women, age ≥18 years old.
* Subject must be a recipient of a non-combined renal transplant from a deceased or living donor. It can be a re transplantation after a graft loss of function or graft rejection
* Subject is willing and able to provide signed written informed consent and willing to comply with study procedures
* Women of Childbearing Potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Subjects who are legally detained in an official institution or under legal protection
* Any condition that, in the opinion of the investigator, might interfere with the patient 's participation in the study, poses an added risk for the patient, or confounds the assessment of the patient
* History of multi-organ transplant (interference with rejection natural history).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
compare levels of eGFR measured by CKD-EPI equation in both arms | 18 months
  Comparison of the levels of eGFR (mL/min/1.73m2) in both arms estimated by glomerular filtration rate (CKD-EPI eGFR) at 18 months' post-transplantation

SECONDARY OUTCOMES:
modification of the immunosuppression treatment | 18 months
  To assess the rate of modification of the immunosuppression treatment in both groups
graft survival rates | 18 months
  To assess predicted graft survival rates in both groups using the iBox
biopsy-proven rejections | 18 months
  compare the rate of biopsy-proven rejections in both groups
incidence of death | 18 months
  compare the incidence of death and allograft loss in both groups
probability of kidney allograft rejection measured by gene expression in the biopsy tissue | 18 months
  determine the probability of different types of rejection (ABMR, TCMR, IFTA and Banff lesions) in kidney transplant recipients' biopsies using gene expression (variance explanation modelling);
quantity of lesion patterns between both groups | 18 months
  identify and compare lesion patterns imaging that are associated with response to rejection therapy using Digital Pathology (immunosuppression dose and response).
compare health care expenses between both groups | 18 months
  compare the cost/benefit of implementing dd-cfDNA monitoring compared to follow-up with the biopsy using the French health insurance database, evaluated at 18 months after transplantation.
compare EQ-5D-5L questionnaire answers between both group | 18 months
  compare the evolution of patient's well-being during the first 18 months after kidney transplantation using the EQ-5D-5L descriptive system and visual analog scale (VAS).
compare the PREMs questionnaire answer in dd-cfDNA-guided group | 18 months
  Level of patient's understanding of their care with non-invasive monitoring and level of satisfaction with it (categorical scale answers from 0 up to 5)
compare the Generalised Anxiety Disorder Assessment (GAD-7 ) questionnaire answer between both group | 18 months
  compare the evolution of patient's well-being during the first 18 months after kidney
compare the visual analyse scale ( VAS ) questionnaire answer between both group | 18 months
  compare the evolution of patient's well-being during the first 18 months after kidney

OTHER OUTCOMES:
rate of biopsies | 18 months
  Comparison of The mean eGFR in both Groups estimated by glomerular filtration rate (CKD-EPI eGFR) at 12 months' post-transplantation and of the number of allograft rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, PR, Study Director — APHP
Locations (6):
- France (6):
  - Georges Pompidou European Hospital, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - AP-HP - Hôpital Tenon, Paris
  - CHU Toulouse, Toulouse
  - Hopital Saint Louis, Paris, Île-de-France Region
  - Hôpital de la Salpêtrière hôpital à Paris, Paris, Île-de-France Region